CLINICAL TRIAL: NCT02500394
Title: Biomarker Guided Intervention to Prevent Development of Acute Kidney Injury in High-risk Surgical Patients
Brief Title: Biomarker Guided Intervention for Prevention of Acute Kidney Injury
Acronym: BigpAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Tobias, Bergler, MD, PD Dr Tobias Bergler, MD, University Hospital Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1476-Version 6
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Acute Kidney Injury
Keywords: renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard care (Placebo Comparator): Patients in the standard care population receive - if biomarkers are elevated -treatment of AKI in accordance with KDIGO 2012 guidelines
  Interventions: Procedure: Ionosteril
- interventional care (Active Comparator): Patients in the interventional population receive - if biomarkers are elevated - individualized treatment/volume substitution (balanced electrolyte solution = Ionosteril; 1,25-5 ml/kg/bw/6 hours) ) on the basis of predefined criteria
  Interventions: Procedure: Ionosteril

INTERVENTIONS:
Procedure: Ionosteril — biomarker guided volume substitution with Ionosteril

SUMMARY:
This study evaluates the impact of a biomarked guided intervention on the development of acute kidney injury in high risk surgical patients. Eligible patients are screened for marker of tubular stress in the urine; if patient specific results are above a pre-defined cutoff they are randomized into a standard care group or an interventional group in which patients receive intensified volume therapy.

DETAILED DESCRIPTION:
This study evaluates the impact of a biomarked guided intervention on the development of acute kidney injury in high risk surgical patients.Used markers have been identified as markers of tubular stress and have been validated in previous studies with more than 1500 patients. The advantage of a biomarker guided approach is the saving of time for the diagnosis a developing acute kidney injury (AKI) in high risk surgical patients, since clinical signs of AKI (rise in creatinine/decline of estimated Glomerular Filtration Rate (eGFR), decline of diuresis). If used biomarkers are above a predefined cutoff within < 4 hours after surgery, patients are randomized in to a standard care population receiving treatment in accordance with Kidney Disease Improving Global Outcomes (KDIGO) guidelines. In the intervention population patients receive individual volume therapy (= balanced electrolyte solution (Ionosteril)) (1,25 ml/kg bw up to 5 ml/kg bw for 6 hours). Degree of volume therapy is estimated by several predifined parameters, e.g. central venous pressure (CVP).

ELIGIBILITY:
"Inclusion Criteria":

* major surgery with a duration > 4 hours plus one of the following criteria:
* age > 75 years, or
* sepsis, or
* shock, or
* polytrauma, or
* need for invasive ventilation or catecholamines, or
* intra-operative application of contrast-medium, or
* preexisting chronic kidney disease (CKD1-4),
* informed consent

Exclusion Criteria:

* age < 18 years,
* end stage renal disease (ESRD),
* preexisting dialysis,
* withdrawal of consent,
* pregnancy,
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AKI in both group | 90 days
  incidence and severity of AKI according to AKI network definition within 90 days will be monitored

SECONDARY OUTCOMES:
need for renal replacement therapy, | 90 days
  Number of participants with a need for renal replacement therapy (defined as dialysis within 90 days)
length of ICU stay | 90 days
  overall length of ICU stay
length of hospital stay | 90 days
  overall length of ICU stay
ICU and hospital costs | 90 days
  to account for resulting costs, ICU and hospital cost of the standard care and the interventional patient population are monitored
incidence of chronic kidney disease (CKD) | 90 days
  Investigators want to see if there are any differences on resulting renal function - different stages of chronic kidney disease (CKD I-V) as a consequence of the performed therapy: standard care accoring to KDIGO guidelines versus interventional care
death | 90 days
  overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Bergler, MD, Principal Investigator — UKR-Department of Nephrology; Ivan Göcze, MD, Principal Investigator — UKR-Department of Surgery
Locations (1):
- University Hospital Center Regensburg, Regensburg, Germany